CLINICAL TRIAL: NCT05152017
Title: Phase I Simple Blind, Placebo Controlled, Randomized Safety and Reactogenicity Trial of the Flu-M Quadro Tetravalent Inactivated Split Influenza Vaccine, Solution for Intramuscular Injection, Produced by FSUE SPbSRIVS FMBA, vs. Placebo in Healthy Volunteers
Brief Title: The Objectives of This Study Are Study the Safety, Reactogenicity and Obtain Preliminary Data on the Immunogenicity of Flu-M Quadro, 4-valent Inactivated Split Influenza Vaccine, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMVq-I-001/18
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-11

CONDITIONS: Influenza
Keywords: influenza; flu; vaccine; Flu-M; FluM Tetra; Tetra; SPbSRIVS; Quadro
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flu-M Quadro with preservative (Experimental): 25 volunteers were vaccinated with the Flu-M Quadro inactivated split influenza vaccine with a preservative
  Interventions: Biological: Flu-M Quadro [inactivated split influenza vaccine] with preservative
- Flu-M Quadro without preservative (Experimental): 25 volunteers were vaccinated with the Flu-M Quadro inactivated split influenza vaccine without a preservative
  Interventions: Biological: Flu-M Quadro [inactivated split influenza vaccine] without preservative
- Placebo (Placebo Comparator): 25 volunteers were vaccinated with a Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Flu-M Quadro [inactivated split influenza vaccine] with preservative — solution for intramuscular injection, 0.5 ml
  Arms: Flu-M Quadro with preservative
Biological: Flu-M Quadro [inactivated split influenza vaccine] without preservative — solution for intramuscular injection, 0.5 ml
  Arms: Flu-M Quadro without preservative
Biological: Placebo — solution for intramuscular injection, 0.5 ml
  Arms: Placebo

SUMMARY:
The study the safety, reactogenicity and obtain preliminary data on the immunogenicity of Flu-M Quadro, 4-valent inactivated split influenza vaccine, in healthy volunteers

DETAILED DESCRIPTION:
The maximum period of the volunteers' participation in the trial will be 35 ± 2 days. Screening period - up to 7 days. The vaccine administration period is 1 day. Follow-up period - 28±2 days.

All volunteers are followed by a clinical investigator for 6 months after vaccination outside of this trial with the aim of detecting possible late adverse reactions. If a volunteer has any delayed-type reactions, the volunteer will be invited to the clinic for correction of his/her condition.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily and personally signed form of informed consent for participation in the trial, before any trial procedure is carried out.
* Verified diagnosis "healthy", at that the clinical investigator shall confirm the absence of pathology on the part of the main organs and systems, previously conducted standard clinical, laboratory and instrumental studies did not reveal any diseases.
* Age between 18 and 60 years old, inclusively.
* Ability to attend all planned visits and all scheduled procedures and studies.
* Willingness of the volunteers to complete Self-Observation Diaries in between their visits to a clinical center.
* Previous vaccination against seasonal influenza at least 9 months prior to inclusion in this trial.
* Consent of the volunteers to use effective contraception methods contraception throughout the trial, including the term of observation for possible post-vaccination reactions

Exclusion Criteria:

* Known hypersensitivity to any of the components of the tested products, as well as to chicken meat or chicken/quail eggs.
* Allergic reaction to any previous influenza vaccination.
* Adverse reaction of severe degree of manifestation or serious adverse reaction to previous influenza vaccine administration.
* Signs of any disease at the time of inclusion in the trial or if less than 4 weeks have expired after recovery.
* Any acute respiratory disease less than 3 months before inclusion in the trial.
* Guillain-Barré syndrome (acute polyneuropathy) in the medical history.
* History of leukemia, tuberculosis, cancer, autoimmune diseases.
* Volunteers who received immunoglobulin or blood products within the last three months before the trial.
* Long-term use (exceeding 14 days) of immunosuppressants, systemic corticosteroids or immunomodulatory agents within 6 months before the trial
* Vaccination with any vaccine within one month before the vaccination.
* Acute infectious or non-communicable diseases, acute exacerbation of a chronic diseases within 4 weeks before the screening.
* Scheduled use of vaccines not provided by the tested protocol within 30 days (inclusively) after the vaccination.
* Pregnant and breastfeeding women.
* Positive blood test results for HIV, syphilis, hepatitis B/C.
* Participation in another clinical trial within 30 days before the screening visit or in parallel with the current trial.
* History of alcohol addiction, drug addiction or abuse of pharmaceutical products.
* Inability or inability to meet the requirements of the protocol, inter lia, for physical, mental or social reasons, according to the clinical investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-11-16 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (local and systemic post-vaccination reactions) | days 1-7
Incidence of adverse events (systemic post-vaccination reactions) | days 1-7
Incidence of any serious adverse events during the trial | days 1-28

SECONDARY OUTCOMES:
The content of specific anti-influenza antibodies in serum | days 0, 28 after the vaccination
The geometric mean titer (GMT) of antibodies to hemagglutinins of the influenza virus | days 0, 28 after the vaccination
Seroconversion factor | days 0, 28
  It shout be more than 2.5 after the vaccination
Seroconversion level | days 0, 28 after the vaccination
Seroprotection level | days 0, 28 after the vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Federally Funded Healthcare Institution Primary Healthcare Unit No. 163, Novosibirsk, Russia